CLINICAL TRIAL: NCT06151197
Title: A Phase 3, Double-blind, Randomized, Placebo-controlled Study to Assess the Efficacy, Safety, and Tolerability of EN3835 vs Placebo in the Treatment of Plantar Fibromatosis (PFI) (Also Known as Ledderhose Disease)
Brief Title: Study to Assess EN3835 in the Treatment of Plantar Fibromatosis (Also Known as Ledderhose Disease)
Acronym: STRIDE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EN3835-309
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Plantar Fibromatosis; Ledderhose Disease
MeSH Terms: conditions — Fibromatosis, Plantar

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EN3835 (Experimental)
  Interventions: Biological: EN3835
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: EN3835 — Biologic: EN3835 injection
  Arms: EN3835
Other: Placebo — Placebo injection
  Arms: Placebo

SUMMARY:
This study will assess the efficacy, safety, and tolerability of EN3835 compared to placebo in the treatment of PFI (also known as Ledderhose disease).

ELIGIBILITY:
Key Inclusion Criteria:

* Be an ambulatory male or female ≥18 years of age.
* Have a diagnosis of PFI.
* Have current foot pain due to PFI.
* Agree not to use prohibited medication, throughout the study, and not use any medication to treat PFI pain, except as permitted per the protocol.
* If female, be of non-childbearing potential (history of hysterectomy, bilateral oophorectomy, bilateral tubal ligation, or postmenopausal with no history of menstrual flow in the 12 months prior to the Screening Visit); or, if of childbearing potential, be non-pregnant, non-lactating and agree to use effective contraception when with a male partner for the duration of the study and for 28 days after any active treatment period.
* Be capable of providing consent, are adequately informed, and understand the nature and risks of the study.

Key Exclusion Criteria:

* Has the presence of non-PFI-related nodules on the foot (for example, neurofibroma, rhabdomyosarcoma, liposarcoma, neurilemmomas, rheumatoid nodules, desmoid tumors, or malignant soft tissue lesions of the foot or ankle).
* Has any musculoskeletal, neuromuscular, neurosensory, other neurological or related disorder that affects the participant's use of his or her foot and/or would impair his/her completion of study assessments as determined by the investigator.
* Has any significant medical history or examination findings related to the participant's plantar nodule(s), which in the investigator's opinion, would make the participant unsuitable for study intervention administration or required assessments and evaluations.
* Has a known bleeding disorder which would make the participant unsuitable for enrollment in the study.
* Has a clinically significant laboratory abnormality.
* Has concurrent diseases that might interfere with the conduct of the study, confound the interpretation of the study results or endanger the participant's well-being, or any significant hematological, endocrine, cardiovascular, respiratory, renal, hepatic, or gastrointestinal disease. If there is a history of such disease but the condition has been stable for greater than 1 year and is judged by the investigator not to interfere with participation in the study, the participant may be included, with the documented approval of the medical monitor.
* Has any other significant medical condition(s), which in the investigator's opinion, would make the participant unsuitable for enrollment in the study.
* Is pregnant or plans to become pregnant.
* Is breastfeeding or is providing or plans to provide breast milk in any manner during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Week 12 in the Weekly Mean of the Average Daily (24-hour) Pain (ADP) Score as Measured on the Pain Intensity Numeric Rating Scale (NRS) | Baseline, Week 12

SECONDARY OUTCOMES:
Change from Baseline in the Foot Function Index (FFI) Difficulty Subscale Score | Baseline, up to Day 85
Change from Baseline in the FFI Activity Limitation Subscale Score | Baseline, up to Day 85
Change from Baseline in the FFI Pain Subscale Score | Baseline, up to Day 85
Change from Baseline in the FFI Total Score | Baseline, up to Day 85
Number of Participants That Used Rescue Analgesic Medication | Up to Day 85
Amount of (milligrams [mg]) Rescue Analgesic Medication Used | Up to Day 85
Patient Global Impression of Change (PGIC) Foot Pain Score | Up to Day 85
Clinician Global Impression of Change (CGIC) Score | Up to Day 85
Subject Satisfaction Score | Up to Day 85
Change from Baseline in Nodule Consistency (Firmness) | Baseline, up to Day 85
Change from Baseline in the Nodular Hardness of the Treated Nodules | Up to Day 85

CONTACTS AND LOCATIONS:
Overall Officials: Luis Ortega, Study Director — Endo Pharmaceuticals
Locations (70):
- United States (63):
  - Endo Site 42, Mesa, Arizona
  - Endo Site 64, Scottsdale, Arizona
  - Endo Site 11, Tucson, Arizona
  - Endo Site 49, Castro Valley, California
  - Endo Site 39, Cerritos, California
  - Endo Site 31, Corona, California
  - Endo Clinical Site 2, Encinitas, California
  - Endo Site 8, Fresno, California
  - Endo Site 28, Lancaster, California
  - Endo Site 9, Los Angeles, California
  - Endo Site 53, Los Angeles, California
  - Endo Site 50, San Francisco, California
  - Endo Site 29, Tarzana, California
  - Endo Site 30, Tarzana, California
  - Endo Site 61, Torrance, California
  - Endo Site 47, Johnstown, Colorado
  - Endo Site 65, Parker, Colorado
  - Endo Site 17, Westminster, Colorado
  - Endo Site 22, Hialeah, Florida
  - Endo Site 59, Jacksonville, Florida
  - Endo Site 33, Medley, Florida
  - Endo Site 23, Miami, Florida
  - Endo Site 21, Miami, Florida
  - Endo Site 35, North Miami Beach, Florida
  - Endo Site 19, Palm Beach Gardens, Florida
  - Endo Clinical Site 1, Pinellas Park, Florida
  - Endo Site 14, Plantation, Florida
  - Endo Site 26, South Miami, Florida
  - Endo Site 60, Sweetwater, Florida
  - Endo Site 24, Lawrenceville, Georgia
  - Endo Site 27, O'Fallon, Illinois
  - Endo Site 45, Oak Brook, Illinois
  - Endo Site 54, Overland Park, Kansas
  - Endo Site 56, Shreveport, Louisiana
  - Endo Site 5, Pasadena, Maryland
  - Endo Site 16, Grand Rapids, Michigan
  - Endo Site 12, Jefferson City, Missouri
  - Endo Site 51, Billings, Montana
  - Endo Site 36, Missoula, Montana
  - Endo Site 34, Oradell, New Jersey
  - Endo Site 62, Vineland, New Jersey
  - Endo Site 15, Durham, North Carolina
  - Endo Site 20, Wilmington, North Carolina
  - Endo Site 63, Oklahoma City, Oklahoma
  - Endo Site 10, Altoona, Pennsylvania
  - Endo Site 44, Malvern, Pennsylvania
  - Endo Site 38, State College, Pennsylvania
  - Endo Site 48, Arlington, Texas
  - Endo Site 3, Bedford, Texas
  - Endo Site 43, Burleson, Texas
  - Endo Site 25, Dallas, Texas
  - Endo Site32, Fort Worth, Texas
  - Endo Site 7, Georgetown, Texas
  - Endo Site 55, Houston, Texas
  - Endo Site 40, Humble, Texas
  - Endo Site 4, McAllen, Texas
  - Endo Site 46, San Antonio, Texas
  - Endo Site 18, San Antonio, Texas
  - Endo Site 37, San Antonio, Texas
  - Endo Site 41, Bountiful, Utah
  - Endo Site 6, Salt Lake City, Utah
  - Endo Site 52, Falls Church, Virginia
  - Endo Site 13, Suffolk, Virginia
- Australia (4):
  - Endo Site 58, East Maitland, New South Wales
  - Endo Site 57, Hunter, New South Wales
  - Endo Site 67, Auchenflower, Queensland
  - Endo Site 66, Victoria Park, Western Australia
- Puerto Rico (3):
  - Endo Site 68, Mayagüez
  - Endo Site 70, Mayagüez
  - Endo Site 69, Ponce

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP